CLINICAL TRIAL: NCT02567149
Title: Intralesional Cidofovir for the Treatment of Recalcitrant Warts in the Pediatric Immune-suppressed Population.
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No funding
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Version 1.0
Record Dates: First submitted 2015-09-30; First posted 2015-10-02 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Warts
Keywords: Wart
MeSH Terms: conditions — Warts | interventions — Cidofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cidofovir (Experimental): Cidofovir clinical resolution of treated warts as evaluated by the investigators
  Interventions: Drug: Cidofovir

INTERVENTIONS:
Drug: Cidofovir — Cidofovir

SUMMARY:
The primary objective is to determine whether intralesional cidofovir is effective at bringing about the total or near-total resolution of warts that have already proven recalcitrant to standard therapy.

The secondary objective is to determine the tolerability of this new mode of administration of cidofovir in the pediatric population

DETAILED DESCRIPTION:
This study includes pediatric patients with history of either primary or iatrogenic immune-suppression who are seeking treatment of warts that have already proven recalcitrant to standard therapy. The first cohort will include 4 patients ages 12 to 17. After all tests indicate treatment safety, the second cohort will be recruited and will include patients ages 8 to 17.

ELIGIBILITY:
Inclusion Criteria:

* 1. The first cohort will include a total of 4 patients ages 12 to 17. After all tests indicate treatment safety, the second cohort will be recruited and will include patients ages 8 to 17.Patient is in immune-suppressed status by one of the following:

  1. Primary immunodeficiency, which may include but is not limited to the following:

     1. Chronic Granulomatous Disease (CGD)
     2. Common Variable Immunodeficiency (CVID)
     3. DiGeorge Syndrome (DGS)
     4. Selective IgA Deficiency
     5. Severe Combined Immunodeficiency (SCID)
     6. X-Linked Agammaglobulinemia (XLA)
  2. Pharmacologic immune-suppressed status from medications including but not limited to:

     1. prednisone
     2. cyclosporine
     3. azathioprine
     4. tacrolimus/ FK506
     5. mycophenolate mofetil
     6. sirolimus

     2. Patient has history of clinically-significant warts that are either refractory to standard therapy or for which standard therapy is contra-indicated or unreasonable 3. Patient has a total wart burden of at least 1cm 4. Patients must have tried and failed at least 2 other conventional treatments for cutaneous warts, including but not limited to:
     * cryotherapy
     * topical salicylic acid
     * imiquimod
     * topical 5FU
     * pulsed dye laser therapy
     * sinecatechins
     * tretinoin or other topical retinoid
     * intralesional candida injection
     * bleomycin
     * electrocautery
     * topical cidofovir cream or gel

     There will be a one month washout period for all treatment modalities, with the exception of intralesional candida, which will be 3 months.

     5. Patient desires ongoing treatment of their warts 6. Patient and/or their parent/guardian consents to participating in this study

     Exclusion Criteria:

  <!-- -->

  1. Treatment area is either ulcerated, secondarily infected, or significantly inflamed
  2. Treatment area is on face or groin area
  3. Patient is pregnant, attempting to become pregnant, or lactating
  4. Patient reports active kidney disease, or chart review reveals recent serum creatinine ≥1.5mg/dL or a history of renal disease/insufficiency or history of diabetes
  5. Patient is currently receiving a nephrotoxic medication
  6. Patient has history of hypersensitivity to cidofovir
  7. Patient is severely ill and/or hospitalized
  8. Patient is receiving chemotherapy

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Clinical resolution of treated warts as evaluated by the investigators | 6 months
  Total or near-total clinical resolution of treated warts as evaluated by the investigators
Improvement of wart-associated symptoms | 6 months
  2. Patient-perceived improvement of wart-associated symptoms

SECONDARY OUTCOMES:
Patient/parent reported tolerability of the treatment | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Polcari, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Medical Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No